CLINICAL TRIAL: NCT00703534
Title: Validation of Patient-reported Outcomes Measures for the Assessment of GERD Symptoms and Their Subsequent Impact on Patients With Partial Response to Proton Pump Inhibitor (PPI) Treatment in a Two Part Multi-center Phase IIa Study Including a Four Week Randomised, Double-blind, Placebo-controlled, Parallel-group Treatment Period
Brief Title: Validation of Patient-reported Outcomes Measures for the Assessment of Gastroesophageal Reflux Disease (GERD) Symptoms
Acronym: C27
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Debra Silberg, MD, Director of Clinical Research, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D9120C00027
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-05

CONDITIONS: GERD; Acid Reflux Disease; Heartburn; Regurgitation
Keywords: GERD; Acid Reflux; Heartburn; Regurgitation; non-acid reflux; PRO measures
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — lesogaberan; Gelusil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD3355 (Experimental)
  Interventions: Drug: AZD3355; Drug: Gelusil®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Gelusil®

INTERVENTIONS:
Drug: AZD3355 — Immediate Release capsule administered as a single dose, 65mg, twice daily for 4 weeks
  Other Names: Lesogaberan
  Arms: AZD3355
Drug: Placebo — capsule. administered as a single dose twice daily for 4 weeks
  Arms: Placebo
Drug: Gelusil® — Chewable tablets taken as needed

SUMMARY:
This research study is being done to gather information about how to do further clinical studies using AZD3355 as an add-on treatment to proton pump inhibitors (PPI).

ELIGIBILITY:
Inclusion Criteria:

* Subject able to read and write US english and able to use electronic devices
* Subjects who have experienced GERD symptoms for at least six months
* Subjects currently taking a prescription or over-the-counter PPI medications for GERD
* Body Mass Index (BMI) 18.5-35.0, inclusive

Exclusion Criteria:

* Subjects that have not experienced any GERD symptoms improvement at all after PPI treatment
* Subjects who have any of the following conditions or diseases- Heart disease, Angina, Seizure disorders such as epilepsy, Congestive Heart Failure (CHF), Liver disease such as Cirrhosis or Hepatitis, Kidney disease, Lung disease or lung cancer, Cancer
* Prior surgery of the upper Gastrointestinal (GI) tract

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Silberg, MD, Study Director — AstraZeneca; Nimish Vakil, MD, Principal Investigator — Aurora Health Center/Waukesha
Locations (84):
- United States (84):
  - Research Site, Athens, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Monterey, California
  - Research Site, Murrieta, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Pueblo, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, DeLand, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Arkansas City, Kansas
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Madisonville, Kentucky
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Elkridge, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Biloxi, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Harrisburg, North Carolina
  - Research Site, Morgantown, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Cranston, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Christiansburg, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Waukesha, Wisconsin
  - Research Site, West End, Wisconsin

REFERENCES:
- [Derived] Ryden A, Leavy OC, Halling K, Stone AA. Comparison of Daily versus Weekly Recording of Gastroesophageal Reflux Disease Symptoms in Patients with a Partial Response to Proton Pump Inhibitor Therapy. Value Health. 2016 Sep-Oct;19(6):829-833. doi: 10.1016/j.jval.2016.05.007. Epub 2016 Jun 29. PMID 27712711
- [Derived] Vakil N, Niklasson A, Denison H, Ryden A. Symptom profile in partial responders to a proton pump inhibitor compared with treatment-naive patients with gastroesophageal reflux disease: a post hoc analysis of two study populations. BMC Gastroenterol. 2014 Oct 10;14:177. doi: 10.1186/1471-230X-14-177. PMID 25304129
- [Derived] Ryden A, Denison H, Karlsson M, Vakil N. Development and validation of a patient-reported outcome instrument in partial responders to proton pump inhibitors. Scand J Gastroenterol. 2013 Sep;48(9):1018-26. doi: 10.3109/00365521.2013.822544. Epub 2013 Aug 6. PMID 23919738

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD3355: AZD3355 capsules 65 mg twice daily, Gelusil tablets as rescue medication if needed
- Placebo: Placebo capsules twice daily, Gelusil tablets as rescue medication if needed
Period: Overall Study
Arm/Group | AZD3355 | Placebo
Started | 235 | 243
Completed | 205 | 218
Not Completed | 30 | 25
Not completed — Adverse Event | 14 | 3
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Incorrect Enrollment | 6 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Severe Non Compliance | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3355 | Placebo | Total
Number analyzed (Participants) | 235 | 243 | 478
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (10.09) | 47.8 (11.5) | 48.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 135 | 280
  Male | 90 | 108 | 198

OUTCOME MEASURES:

1. Primary Outcome: Symptom Intensity Rated by Participants Twice Daily Using an Electronic Reflux Symptom Questionnaire Diary
Description: Symptom intensity rated on a six-graded Likert scale (Did not have; Very mild; Mild; Moderate; Moderately severe; Severe)
Time Frame: Run-in period of 8-12 days and treatment period of 26-30 days
Population: None of the analyses addressing the objectives related to validation of the patient reported outcome measures were made per treatment arm and can therefore not be reported in this format.
Measure: Number; unit: participants
Arm/Group | AZD3355 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | AZD3355 | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 18 | 7
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD3355 | Placebo
Operative Hemorrhage (Injury, poisoning and procedural complications) | 1/235 | 0/243
Suicide Attemp (Psychiatric disorders) | 0/235 | 1/243
Myocardial Infarction (Cardiac disorders) | 0/235 | 1/243
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0/235 | 1/243
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0/235 | 1/243
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD3355 | Placebo
Diarrhoea (Gastrointestinal disorders) | 18/235 | 7/243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AZ shall have 30 days from the proposed final manuscript for any disclosure to review it and may within such time require that submission for publication/disclosure be delayed in order for AZ to file patent applications. If study site/investigator requests permission to publish data(incl oral presentations) it is to be agreed with AZ prior to publ.